CLINICAL TRIAL: NCT05871892
Title: Clinical Impact of 18F-FDGal PET/CT and PET/MRI in Patients Suspected of or Diagnosed With Hepatocellular Carcinoma
Brief Title: 18F-FDGal PET/CT and PET/MRI in Patients With Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-10-72-71-22
Record Dates: First submitted 2023-05-15; First posted 2023-05-23 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-FDGal PET/CT or PET/MRI (Other): Diagnostic scan.
  Interventions: Diagnostic Test: 18F-FDGal PET/CT or PET/MRI

INTERVENTIONS:
Diagnostic Test: 18F-FDGal PET/CT or PET/MRI — All patients suspected of or diagnosed with HCC will be offered an initial 18F-FDGal PET/CT or PET/MRI scan. Moreover, patients who undergo loco-regional treatment (resection, ablation (radiation or microwave), chemo- or radio-embolization) are re-examined with 18F-FDGal. The scans will be performed 1-2 months and 3-5 months after the loco-regional treatment. The images will be analyzed by an experienced PET specialist and the CT or MR images by an experienced radiologist for focal lesions and compared to other imaging modalities. The investigators expect approximately 25 patients per year during a 5-year period and as such aim at a total of 125 patients

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common primary liver tumor and the fourth leading cause of cancer-related death worldwide. In Denmark, the incidence of HCC is 5.2 per 100.000 population per year with a dismal prognosis as the median survival time is just 7.7 months.

Extrahepatic spread of HCC is common at advanced stages with haematogenous spread to lungs, bones and adrenal glands or lymphatic spread to regional lymph nodes.

The majority of patients who develop HCC have cirrhosis of the liver and in these patients, diagnosis can be made non-invasively with characteristic contrast-enhancement pattern on computed tomography (CT) and/or magnetic resonance imaging (MRI). Although contrast-enhanced CT and MRI are considered equal in current guidelines, MRI may have a better sensitivity especially for small lesions.

Positron emission tomography (PET) is a molecular imaging technique based on the injection of a very small dose of a tracer substance labelled with a positron emitting radioisotope. PET with the glucose tracer 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (18F-FDG) is an important tool in the staging of many cancer forms, but it is not included in the international guidelines for management of HCC because of suboptimal sensitivity of only up to 50-60 % for HCC situated in the liver.

In Aarhus, the liver specific tracer 18F-FDGal has been developed. It is a fluorine-18 labelled galactose analogue which in the human body is trapped in hepatocytes by phosphorylation by galactokinase. The first study of the diagnostic use of 18F-FDGal PET/CT in patients suspected of having HCC was published in 2011. The study showed good clinical potential for 18F-FDGal as a tracer for detection of intra- as well as extrahepatic HCC.

The aim of the present project is to establish the clinical impact and utilization of 18F-FDGal PET/CT and PET/MRI in patients suspected of having HCC or diagnosed with HCC, for staging and evaluation of treatment response including effect of treatment on liver function.

Hypotheses:

I. Adding 18F-FDGal PET/CT or PET/MRI to diagnostic work-up of patients suspected of or diagnosed with HCC will add to the establishment of a definitive diagnosis and improve staging and thus choice of treatment.

II. The uptake pattern of 18F-FDGal in HCC provides prognostic information and can be used to evaluate regional metabolic liver function before and after loco-regional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly-referred patients suspected of or diagnosed with HCC
* Age above 18 years

Exclusion Criteria:

* The patient does not want to take part in the study
* The responsible investigator determines that the patient is not qualified for a PET scan.
* Patients who are offered systemic chemotherapy or best supportive care will be excluded.
* Renal insufficiency (estimated glomerular filtration rate [eGFR] <30 ml/min/1.73 m2 body surface area).
* Pregnant or nursing patients.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the PET tracer 18F-FDGal | Five years
  The ability of the scan 18F-FDGal PET/CT or PET/MRI to correctly identify lesions representing intrahepatic and/or extrahepatic hepatocellular carcinoma.
Metabolic function of the liver evaluated by the PET tracer 18F-FDGal | Five years
  The ability of the scan 18F-FDGal PET/CT or PET/MRI to determine the loco-regional treatment effects on metabolic liver function in other regions of the liver.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No